CLINICAL TRIAL: NCT05028816
Title: Force Modulating Tissue Bridges for Closure of Vertical Scars in Breast Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey M. Kenkel, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: STU 2021-0791
Record Dates: First submitted 2021-08-27; First posted 2021-08-31 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Surgical Incision
Keywords: Wound Healing
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Intervention Model Description: Randomization will occur after all the portions of the surgical procedure are completed except for final skin layer closure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be unknown to PI and additional care providers until an envelope is opened by research staff at the time of final layer closure in the OR.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (Other): Side 1: Final layer dermal closure with poliglecaprone 25 suture (Monocryl ®, Ethicon, Inc. Bridgewater, NJ)
  Side 2: Final layer closure with force modulating tissue bridges (FMTB) (Brijjit BP100-6, Brijjit Medical Inc., Marietta, GA)
  Interventions: Other: Side 1: Final layer dermal closure with poliglecaprone 25 suture; Device: Side 2: Final layer closure with force modulating tissue bridges (FMTB)
- Group 2 (Other): Side 1: Final layer closure with force modulating tissue bridges (FMTB) (Brijjit BP100-6, Brijjit Medical Inc., Marietta, GA)
  Side 2: Final layer dermal closure with poliglecaprone 25 suture (Monocryl ®, Ethicon, Inc. Bridgewater, NJ)
  Interventions: Device: Side 1: Final layer closure with force modulating tissue bridges (FMTB); Other: Side 2: Final layer dermal closure with poliglecaprone 25 suture

INTERVENTIONS:
Device: Side 1: Final layer closure with force modulating tissue bridges (FMTB) — Brijjit is a non-invasive wound closure device that reduces tension on scars and aids improving scar appearance.
  Other Names: Brijjit
  Arms: Group 2
Other: Side 1: Final layer dermal closure with poliglecaprone 25 suture — Current method of wound closure
  Arms: Group 1
Device: Side 2: Final layer closure with force modulating tissue bridges (FMTB) — Brijjit is a non-invasive wound closure device that reduces tension on scars and aids improving scar appearance.
  Other Names: Brijjit
  Arms: Group 1
Other: Side 2: Final layer dermal closure with poliglecaprone 25 suture — Current method of wound closure
  Arms: Group 2

SUMMARY:
This is a prospective, within-subject randomized, single blinded study designed to follow up to forty-two (42) qualified and consenting adult females, 18-65 years of age scheduled for elective breast reduction surgery using a standard inverted Wise (inverted "T") incision pattern

DETAILED DESCRIPTION:
This is a prospective, within-subject randomized, single blinded study designed to follow up to forty-two (42) qualified and consenting adult females, 18-65 years of age scheduled for elective breast reduction surgery using a standard inverted Wise (inverted "T") incision pattern. Subjects will be randomized to the method of closure and wound support of the symmetrical vertical breast incisions. On the intervention side subjects will have FMTBs applied for final layer closure of the vertical breast incision and will continue with repeat application every two weeks for ongoing wound support for a total of 8 weeks of therapy. On the control side standard suture closure and wound dressings will be utilized. Patients will be evaluated at two-week intervals up until 8 weeks post-operative, then will have 3 additional follow up visits at 3-months, 6-months and 12-months post-operatively. The effects of the therapy will be analyzed during the follow up visits through photography, skin assessments and POSAS (Patient and Observer Scar Assessment Scale) results. A subgroup of 10 patients will also undergo biopsies of the area of interest at five time points throughout the study. Primary study outcomes include POSAS results and photographic assessment while secondary outcomes include scar volume/surface area, gene regulation and genetic analysis obtained via biopsies, collagen volume, skin assessments, colorimetry and time of length of adherence of the device.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult females 18-65 years of age
2. Planned procedure is bilateral breast reduction with modified Wise (anchor, inverted "T") scar pattern.
3. Ability to adhere wound therapy after surgery for 8 weeks or have a willing family member/partner to assist with wound therapy care.
4. Willing to follow wound care therapy as instructed by study staff.
5. Willing to return for follow up visits and undergo study evaluations.

Exclusion Criteria:

1. Individuals diagnosed with known allergy to general adhesives/adhesive tape
2. Individuals with a history of using the following prescription medications:

   * Accutane within the past year;
   * Systemic steroid use within the past year
3. Individuals who have significant scarring on the test site/area(s)
4. Individuals with malnutrition
5. Individuals who have a body mass index >35
6. Individual who have a history of radiation therapy
7. Individual who have a history of breast cancer
8. Active smokers
9. Individuals with a disorder known to negatively affect wound healing (e.g. autoimmune disease, connective tissue disease
10. Individual who have an observable pre-operative or intra-operative breast asymmetry that, in the investigators opinion, would interfere with the evaluation of the efficacy of the wound therapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 39 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — Chairman, UT Southwestern
Locations (1):
- UT Southwestern Medical Center- Outpatient Building, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FMTB Left/ SOC Right: SOC: Final layer dermal closure with poliglecaprone 25 suture (Monocryl ®, Ethicon, Inc. Bridgewater, NJ)
  Briijt: Final layer closure with force modulating tissue bridges (FMTB) (Brijjit BP100-6, Brijjit Medical Inc., Marietta, GA)
- SOC Left/FMTB Right: SOC: Final layer dermal closure with poliglecaprone 25 suture (Monocryl ®, Ethicon, Inc. Bridgewater, NJ)
  FMTB: Final layer closure with force modulating tissue bridges (FMTB) (Brijjit BP100-6, Brijjit Medical Inc., Marietta, GA)
Period: Overall Study
Arm/Group | FMTB Left/ SOC Right | SOC Left/FMTB Right
Started | 20 | 16
Completed | 10 | 12
Not Completed | 10 | 4
Not completed — Lost to Follow-up | 5 | 3
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Subjects: Subjects consented and treated in the study
Arm/Group | Study Subjects
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS)- Patient Scores 12M
Description: Validated scale used to assess the scar quality after surgery from patient and observer (clinician) prospective.
  Scoring:
  Each of the six items on both the Observer and Patient scales is scored on a 10-point numerical rating scale, where:
  1 represents tissue that is like normal skin. 10 represents the worst scar imaginable for the observer, or the worst imaginable sensation/difference for the patient.
  The total score for each scale is the sum of the scores for the six items, ranging from 6 to 60. A higher score indicates a poorer scar quality while a lower scores indicates an ideal scar outcome.
Time Frame: 12 Months
Population: All subjects received an FTMB and SOC closure on either surgical scar
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- FTMB Scar: Subjects assessed the scar treated with FTMB
- SOC Scar: Subjects assessed scars closed with standard care closure
Arm/Group | FTMB Scar | SOC Scar
Number analyzed (Participants) | 23 | 20
score on a scale
  Pain | 1.09 (0.42) | 1.22 (0.74)
  Itchiness | 1.3 (1.06) | 1.87 (1.96)
  Color | 4.22 (2.92) | 1.22 (0.74)
  Stiffness | 2.17 (1.61) | 2.39 (1.99)
  Thickness | 2.74 (2.03) | 2.74 (2.22)
  Irregularities | 2.70 (1.61) | 2.70 (1.87)
  Total Score | 14.22 (7.25) | 15.22 (8.63)
  Overall Opinion | 3.17 (1.87) | 3.04 (2.14)

2. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS)- Patient Scores 6M
Description: as for outcome 1
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FTMB Scar | SOC Scar
Number analyzed (Participants) | 20 | 20
score on a scale
  Pain | 1.05 (0.23) | 1.00 (0)
  Itchiness | 1.11 (0.32) | 1.22 (0.55)
  Color | 4.37 (2.67) | 4.53 (2.99)
  Stiffness | 3.32 (2.43) | 3.32 (2.24)
  Thickness | 3.95 (2.66) | 3.58 (2.73)
  Irregularity | 4.16 (2.67) | 3.95 (2.72)
  Total score | 17.95 (9.73) | 17.53 (9.98)
  Overall Opinion | 3.68 (2.16) | 3.26 (2.02)

3. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS)- Patient Scores 3M
Description: as for outcome 1
Time Frame: 3 Months
Population: All subjects received an FTMB and SOC closure on either surgical scar
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FTMB Scar | SOC Scar
Number analyzed (Participants) | 20 | 20
score on a scale
  Pain | 1.30 (0.8) | 1.30 (0.66)
  Itchiness | 2.40 (2.11) | 2.15 (1.69)
  Color | 4.55 (2.78) | 4.60 (2.85)
  Stiffness | 3.8 (2.97) | 3.75 (2.84)
  Thickness | 3.20 (2.38) | 3.35 (2.66)
  Irregularities | 3.5 (2.4) | 3.45 (2.5)
  Total Score | 18.75 (10.15) | 18.55 (9.94)
  Overall Opinion | 4.15 (2.46) | 4.15 (2.43)

4. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS)- Observer Scores 3M
Description: as for outcome 1
Time Frame: 3 Months
Population: All subjects received an FTMB and SOC closure on either surgical scar
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FTMB Scar | SOC Scar
Number analyzed (Participants) | 20 | 20
score on a scale
  Vascularity | 1.45 (0.76) | 1.70 (0.73)
  Pigmentation | 1.75 (0.97) | 2.20 (1.20)
  Thickness | 1.55 (1) | 1.90 (0.97)
  Relief | 1.40 (0.94) | 1.60 (0.99)
  Pliability | 1.30 (0.92) | 1.50 (0.95)
  Surface Area | 1.30 (0.73) | 1.75 (0.85)

5. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS)- Observer Scores 12M
Description: as for outcome 1
Time Frame: 12 Months
Population: All subjects received an FTMB and SOC closure on either surgical scar
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FTMB Scar | SOC Scar
Number analyzed (Participants) | 23 | 23
score on a scale
  Vascularity | 1.26 (0.45) | 1.30 (0.56)
  Pigmentation | 1.74 (0.81) | 2.04 (0.88)
  Thickness | 1.70 (0.88) | 1.96 (0.77)
  Relief | 1.30 (0.56) | 1.57 (0.79)
  Pliability | 1.35 (0.57) | 1.57 (0.73)
  Surface Area | 1.35 (0.57) | 1.78 (0.85)

6. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS)- Observer Scores 6M
Description: as for outcome 1
Time Frame: 6 Months
Population: All subjects received an FTMB and SOC closure on either surgical scar
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FTMB Scar | SOC Scar
Number analyzed (Participants) | 20 | 20
score on a scale
  Vascularity | 1.47 (0.77) | 1.53 (0.77)
  Pigmentation | 1.68 (0.82) | 2.37 (0.96)
  Thickness | 1.32 (0.48) | 1.63 (0.68)
  Relief | 1.16 (0.69) | 1.32 (0.58)
  Pliability | 1.16 (0.69) | 1.11 (0.46)
  Surface Area | 1.16 (0.37) | 1.26 (0.56)

7. Secondary Outcome: Scar Area Assessment
Description: eKare will be used to asses scars progression over an 8-week period.
  The data is an average at each timepoints.
Time Frame: Week 2, Week 4, Week 6 and Week 8
Measure: Mean (Standard Error); unit: cm^2
Groups:
- FMTB: Closure with FMTB
- Suture: Closure with suture
Arm/Group | FMTB | Suture
Number analyzed (Participants) | 18 | 18
cm^2
  Overall | 1.53 (0.10) | 2.16 (0.11)
  Week 2 | 1.61 (0.14) | 2.28 (0.20)
  Week 4 | 1.69 (0.13) | 2.65 (0.17)
  Week 6 | 1.57 (0.10) | 1.93 (0.25)
  Week 8 | 1.25 (0.17) | 2.63 (0.20)

8. Secondary Outcome: Gene Regulation- Elastin
Description: Assessment of mechanical properties of regenerated skin
  Fold change= sample/average of the baseline
Time Frame: Baseline, 4 Week, 8 Week, 3 Months, 12 Months
Measure: Mean (Standard Error); unit: fold change
Groups:
- FMTB- Baseline; FMTB- Week 4; FMTB- Week 8; FMTB- Month 3; FMTB- Month 12: Subjects with FMTB closure
- Suture- Baseline; Sutures- Week 4; Suture- Week 8; Suture Month 3; Suture- Month 12: Subjects with standard of care closure
Arm/Group | FMTB- Baseline | FMTB- Week 4 | FMTB- Week 8 | FMTB- Month 3 | FMTB- Month 12 | Suture- Baseline | Sutures- Week 4 | Suture- Week 8 | Suture Month 3 | Suture- Month 12
Number analyzed (Participants) | 11 | 6 | 9 | 9 | 5 | 11 | 6 | 9 | 9 | 5
fold change | 1.09 (0.16) | 0.80 (0.09) | 1.04 (0.07) | 0.82 (0.08) | 1.21 (0.33) | 0.92 (0.14) | 1.01 (0.07) | 1.17 (0.09) | 1.21 (0.11) | 1.22 (0.22)

9. Secondary Outcome: Gene Analysis- Macrophage
Description: Biopsy will be obtained to assess progression of tissue Fold change= sample/average of the baseline
Time Frame: Baseline, 4 Week, 8 Week, 3 Months, 12 Months
Measure: Mean (Standard Error); unit: fold change
Arm/Group | FMTB- Baseline | FMTB- Week 4 | FMTB- Week 8 | FMTB- Month 3 | FMTB- Month 12 | Suture- Baseline | Sutures- Week 4 | Suture- Week 8 | Suture Month 3 | Suture- Month 12
Number analyzed (Participants) | 11 | 6 | 9 | 9 | 5 | 11 | 6 | 9 | 9 | 5
fold change | 1.00 (0.18) | 0.77 (0.04) | 0.99 (0.10) | 0.98 (0.22) | 0.50 (0.05) | 1.000 (0.17) | 0.69 (0.14) | 1.07 (0.14) | 0.82 (0.30) | 0.56 (0.04)

10. Secondary Outcome: Histology Collagen 3
Description: Biopsy will be obtained to assess early wound healing and ECM formation during scaffold integration Fold change= sample/average of the baseline
Time Frame: Baseline, 4 Week, 8 Week, 3 Months, 12 Months
Measure: Mean (Standard Error); unit: fold change
Arm/Group | FMTB- Baseline | FMTB- Week 4 | FMTB- Week 8 | FMTB- Month 3 | FMTB- Month 12 | Suture- Baseline | Sutures- Week 4 | Suture- Week 8 | Suture Month 3 | Suture- Month 12
Number analyzed (Participants) | 11 | 6 | 9 | 9 | 5 | 11 | 6 | 9 | 9 | 5
fold change | 1.11 (0.21) | 1.19 (0.22) | 1.13 (0.22) | 1.37 (1.46) | 1.46 (0.11) | 0.89 (0.14) | 0.89 (0.18) | 1.38 (0.22) | 1.13 (0.31) | 1.51 (0.19)

11. Secondary Outcome: Change in Mechanical Properties of Human Tissue
Description: BTC2000 is used to assess changes in skin laxity and elasticity in skin that was treated with each closure. Skin maximum pressure, laxity, elastic/viscoelastic/ultimate deformation, and elasticity is measured to track changes through multiple timepoints.
Time Frame: Baseline, 3 Months, 6 Months, and 12 Months
Population: Analysis by closure and timepoints
Measure: Mean (Standard Deviation); unit: mm
Groups:
- FTMB- Baseline; FTMB- 3M; FTMB- 6M; FTMB- 12M: Subjects with FMTB closure
- SOC- Baseline; SOC- 3M; SOC- 6M; SOC- 12M: Subjects with standard of care closure
Arm/Group | FTMB- Baseline | FTMB- 3M | FTMB- 6M | FTMB- 12M | SOC- Baseline | SOC- 3M | SOC- 6M | SOC- 12M
Number analyzed (Participants) | 23 | 20 | 20 | 23 | 23 | 20 | 20 | 23
mm
  Maximum Pressure (mm) | 149.70 (0.56) | 149.70 (0.47) | 149.58 (0.51) | 149.62 (0.50) | 149.78 (0.42) | 149.70 (0.47) | 149.58 (0.51) | 149.62 (0.50)
  Laxity (mm) | 1.14 (0.60) | 0.98 (0.43) | 1.26 (0.46) | 1.53 (0.59) | 1.13 (0.60) | 1.04 (0.4) | 1.28 (0.39) | 1.53 (0.59)
  Elastic Deformation (mm) | 1.58 (0.63) | 1.56 (0.41) | 1.82 (0.41) | 2.02 (0.58) | 1.62 (0.65) | 1.66 (0.49) | 1.86 (0.38) | 2.07 (0.54)
  Viscoelastin Deformation (mm) | .06 (.02) | .08 (.03) | .08 (.02) | .09 (.03) | .07 (.02) | .08 (.03) | .08 (.02) | .08 (.02)
  Ultimate Deformation (mm) | 1.64 (0.63) | 1.64 (0.41) | 1.91 (0.41) | 2.11 (0.58) | 1.68 (0.67) | 1.74 (0.50) | 1.94 (0.38) | 2.15 (0.54)
  Elasticity (mm) | 0.97 (0.48) | 0.85 (0.26) | 1.07 (0.34) | 1.17 (0.53) | 1.00 (0.52) | 0.89 (0.38) | 1.03 (0.31) | 1.22 (0.43)

12. Secondary Outcome: Histology Collagen 1
Description: Biopsy will be obtained to assess collagen synthesis, restoring dermal strength and elasticity during regeneration fold change= sample/average of the baseline
Time Frame: Baseline, 4 Week, 8 Week, 3 Months, 12 Months
Measure: Mean (Standard Error); unit: fold change
Groups:
- FMTB- Baseline; FMTB- Week 4; FMTB- Week 8; FMTB- Month 3; FMTB- Month 12: Subject received FMTB closure
- Suture- Baseline; Sutures- Week 4; Suture- Week 8; Suture Month 3; Suture- Month 12: Subject received suture closure
Arm/Group | FMTB- Baseline | FMTB- Week 4 | FMTB- Week 8 | FMTB- Month 3 | FMTB- Month 12 | Suture- Baseline | Sutures- Week 4 | Suture- Week 8 | Suture Month 3 | Suture- Month 12
Number analyzed (Participants) | 11 | 6 | 9 | 9 | 5 | 11 | 6 | 9 | 9 | 5
fold change | 1.00 (0.25) | 1.02 (0.13) | 0.92 (0.16) | 1.17 (0.20) | 0.92 (0.15) | 1.00 (0.16) | 0.91 (0.12) | 0.97 (0.17) | 1.18 (0.25) | 1.04 (0.07)

13. Secondary Outcome: Scar Maximum Depth
Description: eKare will be used to asses scar area
Time Frame: Week 2, Week 4, Week 6 and Week 8
Measure: Mean (Standard Error); unit: mm
Arm/Group | FMTB | Suture
Number analyzed (Participants) | 18 | 18
mm
  Overall | 0.07 (0.01) | 0.09 (0.00)
  Week 2 | 0.09 (0.01) | 0.10 (0.00)
  Week 4 | 0.07 (0.02) | 0.09 (0.01)
  Week 6 | 0.08 (0.01) | 0.1 (0.01)
  Week 8 | 0.04 (0.02) | 0.09 (0.02)

14. Secondary Outcome: Interleukin-8 (IL8)
Description: IL8 is a small protein called a chemokine that play a crucial role in the body's immune and inflammatory responses. A biopsy will be obtained at different timepoints to assessment changes from baseline.
  fold change= sample/average of the baseline
Time Frame: Baseline, 4 Week, 8 Week, 3 Months, 12 Months
Measure: Mean (Standard Error); unit: fold change
Arm/Group | FMTB- Baseline | FMTB- Week 4 | FMTB- Week 8 | FMTB- Month 3 | FMTB- Month 12 | Suture- Baseline | Sutures- Week 4 | Suture- Week 8 | Suture Month 3 | Suture- Month 12
Number analyzed (Participants) | 11 | 6 | 9 | 9 | 5 | 11 | 6 | 9 | 9 | 5
fold change | 1.39 (0.51) | 30.49 (11.97) | 14.75 (8.29) | 9.38 (3.26) | 0.18 (0.04) | 1.09 (0.30) | 10.50 (0.58) | 0.41 (0.21) | 13.24 (10.64) | 1.13 (0.42)

15. Secondary Outcome: Interleukin-6 (IL6)
Description: IL6 is an inflammatory cytokineses that measures acute phase response following treatment. A biopsy will be obtained at different timepoints to assessment changes from baseline.
  fold change= sample/average of the baseline
Time Frame: Baseline, 4 Week, 8 Week, 3 Months, 12 Months
Measure: Mean (Standard Error); unit: fold change
Arm/Group | FMTB- Baseline | FMTB- Week 4 | FMTB- Week 8 | FMTB- Month 3 | FMTB- Month 12 | Suture- Baseline | Sutures- Week 4 | Suture- Week 8 | Suture Month 3 | Suture- Month 12
Number analyzed (Participants) | 11 | 6 | 9 | 9 | 5 | 11 | 6 | 9 | 9 | 5
fold change | 1.25 (1.19) | 2.89 (1.40) | 2.23 (1.69) | 7.96 (2.96) | 0.53 (0.15) | 5.89 (3.99) | 2.07 (0.06) | 2.83 (0.85) | 5.24 (1.34) | 1.75 (1.10)

16. Secondary Outcome: Measure of the Skins Function
Description: TEWL is a skin measurement to objectively measure the skins barrier function. The device measures the rate at which water evaporates from the skins surface
Time Frame: Baseline, 3 Months, 6 Months, and 12 Months
Population: Analysis by closure and timepoints
Measure: Mean (Standard Deviation); unit: g/m^2/h
Groups:
- Forced Modulated Tissue Bridges: Subjects with FMTB closure
- Standard of Care: Subjects with standard of care closure
Arm/Group | Forced Modulated Tissue Bridges | Standard of Care
Number analyzed (Participants) | 23 | 23
g/m^2/h
  Baseline | 10.01 (4.77) | 10.45 (6.84)
  3 Months | 10.53 (3.96) | 9.64 (2.92)
  6 Months | 9.97 (2.89) | 9.78 (2.88)
  12 Months | 9.03 (3.53) | 9.56 (3.41)

17. Secondary Outcome: Change in Tissue Density
Description: Epidermal and Dermis density was measured with a high frequency ultrasound to understand the changes to the structure and composition of the skin.
Time Frame: Baseline, 3 Months, 6 Months, and 12 Months
Population: Analysis by closure and timepoints
Measure: Mean (Standard Deviation); unit: g/cm^3
Groups:
- Forced Modulated Tissue Bridges- Epidermis; Forced Modulated Tissue Bridges- Dermis: Subjects with FMTB closure
- Standard of Care- Epidermis; Standard of Care- Dermis: Subjects with standard of care closure
Arm/Group | Forced Modulated Tissue Bridges- Epidermis | Forced Modulated Tissue Bridges- Dermis | Standard of Care- Epidermis | Standard of Care- Dermis
Number analyzed (Participants) | 23 | 20 | 23 | 20
g/cm^3
  Baseline | 81.53 (20.64) | 55.08 (18.40) | 82.67 (22.28) | 53.53 (21.36)
  3 Months | 83.37 (16.38) | 28.92 (10.59) | 83.37 (16.38) | 31.87 (13.17)
  6 Months | 84.33 (21.15) | 23.55 (15.43) | 84.33 (21.15) | 75.02 (9.40)
  12 Months | 78.27 (13.68) | 18.70 (8.82) | 23.50 (14.38) | 20.02 (9.86)

18. Secondary Outcome: Change in Tissue Thickness
Description: Epidermal and Dermis thickness was measured with a high frequency ultrasound to understand the changes to the structure and composition of the skin.
Time Frame: Baseline, 3 Months, 6 Months, and 12 Months
Population: Analysis by closure and timepoints
Measure: Mean (Standard Deviation); unit: um
Arm/Group | Forced Modulated Tissue Bridges- Epidermis | Forced Modulated Tissue Bridges- Dermis | Standard of Care- Epidermis | Standard of Care- Dermis
Number analyzed (Participants) | 23 | 20 | 23 | 20
um
  Baseline | 102.43 (18.70) | 1020.87 (237.74) | 102.91 (197.33) | 977.61 (180.79)
  3 Months | 92.42 (13.31) | 1073.79 (223.75) | 92.42 (13.31) | 1073.79 (223.75)
  6 Months | 96.74 (19.09) | 1118.37 (305.19) | 96.74 (19.09) | 1118.37 (305.19)
  12 Months | 98.90 (15.23) | 1081.14 (321.27) | 150.70 (197.33) | 1915.65 (3568.82)

19. Secondary Outcome: Change in Tissue Stiffness
Description: Tissue stiffness was measured using the BTC2000 to measure the resistance of the tissue under applied force/pressure.
Time Frame: Baseline, 3 Months, 6 Months, and 12 Months
Population: Analysis by closure and timepoints
Measure: Mean (Standard Deviation); unit: mmHg/mm
Arm/Group | Forced Modulated Tissue Bridges | Standard of Care
Number analyzed (Participants) | 23 | 23
mmHg/mm
  Baseline | 232.89 (70.29) | 16991.96 (80448.37)
  3 Months | 179.50 (40.27) | 185.53 (80.62)
  6 Months | 173.03 (19.12) | 166.90 (30.79)
  12 Months | 170.31 (31.14) | 170.23 (30.98)

20. Secondary Outcome: Change in Tissue Energy Absorption
Description: Tissue energy absorption was measured using the BTC2000 to measure the softness of the tissue through the deformation process.
Time Frame: Baseline, 3 Months, 6 Months, and 12 Months
Population: Analysis by closure and timepoints
Measure: Mean (Standard Deviation); unit: mmHg*mm
Arm/Group | Forced Modulated Tissue Bridges | Standard of Care
Number analyzed (Participants) | 23 | 23
mmHg*mm
  Baseline | 66.80 (19.42) | 69.77 (22.87)
  3 Months | 77.17 (15.40) | 81.04 (21.15)
  6 Months | 81.28 (10.19) | 84.57 (13.99)
  12 Months | 85.05 (15.08) | 85.32 (13.80)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- FMTB: Final layer closure with force modulating tissue bridges (FMTB) (Brijjit BP100-6, Brijjit Medical Inc., Marietta, GA)
- Suture: SOC: Final layer dermal closure with poliglecaprone 25 suture (Monocryl ®, Ethicon, Inc. Bridgewater, NJ)
Arm/Group | FMTB | Suture
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/36 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMTB (N=36) | Suture (N=36)
Contact Dermititis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Oral Thrush (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT05028816/Prot_SAP_000.pdf